CLINICAL TRIAL: NCT04768153
Title: Prioritising Prevention of COVID-19 in Persons With Cancer in the French West Indies: Monitoring Psychological Impact to Optimize Healthcare Delivery Strategies in Unique Public Health Circumstances
Brief Title: Prioritising Prevention of COVID-19 in Persons With Cancer in the French West Indies
Acronym: RESILIENCE
Status: Terminated | Type: Observational
Why Stopped: Poor recruitment
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 20_RIPH3_04
Record Dates: First submitted 2021-02-09; First posted 2021-02-24 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Cancer
Keywords: Psychiatry; Public health
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Realization of the COVID -19 serological profile of cancer patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients
  Interventions: Biological: Serology

INTERVENTIONS:
Biological: Serology — Serological diagnosis of COVID-19 in patients with cancer from a sample of cancer patients, at 3 and 6 months after implementation of confinement in France

SUMMARY:
The public health council (Haut Conseil de Santé Publique) published a statement on 14 March 2020 relating to the management of patients with severe forms of COVID-19, stipulating specific recommendations for patients with cancer.

The statement notes that patients with cancer at much higher risk (four to five times higher) of several respiratory complications, which develop very rapidly, especially if they had recently undergone surgery or chemotherapy in the previous few weeks, and that this risk could be life-threatening, on top of the cancer-related risk. In addition, the statement noted that:

* COVID-19 appears to be more frequent in patients with cancer than among the general population (1% vs 0.29%)
* Among those infected, the risk of severe respiratory complications requiring admission to the intensive care unit (ICU) is higher in patients with cancer than among those without (39% vs 8%, P=0.0003).
* A history of chemotherapy or surgery in the previous months is an important prognostic factor for the development of severe respiratory complications (odds ratio (OR) = 5.34, P= 0.0026).
* Deterioration of respiratory function occurs more quickly in patients with cancer (13 vs 43 days, hazard ratio (HR) 3.56, 95% confidence interval (CI) [1.65-7.69]).

In addition, COVID-19 may lead to a change in the diagnostic and therapeutic management of patients with cancer, with potential consequences such as use of oral treatments at home, discontinuation of anticancer therapy depending on the context, or prioritization of management according to curative/palliative treatment type, age, and line of therapy.

International studies previously reported the psychological repercussions of major epidemics on the emotional state. The impact of COVID-19 on patients with cancer therefore warrants evaluation, among cancer patients in the French West Indies, in the current situation of nationwide lockdown.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older living in the French West Indies
* Patient with prevalent cancer of the prostate, breast, lung, colon or rectum
* Patients who receive the information leaflet and do not express any opposition to the use of their personal medical data

Exclusion Criteria:

* Patients who are unable to answer the study questionnaires
* Patients who do not speak fluent French
* Persons under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cancer patients followed at the Martinique University Hospital
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of Psychiatric disorders | 3 months after implementation of confinement in France
  Evaluation of presence of psychiatric disorders by questionnaire after the initiation of population-level confinement due to the COVID-19 epidemic
Evaluation of Psychiatric disorders | 6 months after implementation of confinement in France
  Evaluation of presence of psychiatric disorders by questionnaire after the initiation of population-level confinement due to the COVID-19 epidemic

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No